CLINICAL TRIAL: NCT06164353
Title: Clinical and Radiographic Evaluation of the Peri-implant Tissue Changes Around Early Placed Implants in the Esthetic Zone With Contour Augmentation Using Autogenous Partially Demineralized Dentin Graft Versus Xenograft: A RCT
Brief Title: the Peri-implant Tissue Changes Around Implants in the Esthetic Zone Using Demineralized Dentin Graft vs Xenograft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Saeed Hassan Alqahtani, Principal Investigator Rana Saeed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER6-32
Record Dates: First submitted 2023-11-12; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Implant Site Reaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bovine xenograft covered with a collagen membrane (Active Comparator): The same procedure of implant placement will be performed but xenograft will be used for augmentation.
  In both groups, the placed graft will be covered with a collagen membrane. Finally, tension free wound closure will be attained after periosteal releasing incision and suturing using 5/0 proline interrupted sutures.
  An immediate postoperative CBCT scan will be done following the surgical procedure.
  Interventions: Biological: Partially demineralized dentin graft covered with a collagen membrane
- Partially demineralized dentin graft covered with a collagen membrane (Experimental): The stored tooth will undergo grinding using the tooth transformer device. The produced particulate dentin graft will be of a particle size 400-800 µm. Afterwards, these particles will undergo partial demineralization by immersion in in 2% HNO3 for 10 minutes. Then, it will be washed twice using phosphate buffered saline. The exposed implant threads will be covered by partially demineralized autogenous dentin graft in the test group
  Interventions: Biological: Partially demineralized dentin graft covered with a collagen membrane

INTERVENTIONS:
Biological: Partially demineralized dentin graft covered with a collagen membrane — The stored tooth will undergo grinding using the tooth transformer device. The produced particulate dentin graft will be of a particle size 400-800 µm. Afterwards, these particles will undergo partial demineralization by immersion in in 2% HNO3 for 10 minutes. Then, it will be washed twice using phosphate buffered saline. The exposed implant threads will be covered by partially demineralized autogenous dentin graft in the test group

SUMMARY:
Dentin grafts are categorized into mineralized dentin, partially demineralized dentin matrix (PDDM), and demineralized dentin matrix (DDM). Mineralized dentin can be obtained from a dentin grinder and was found to be less effective in bone formation, while DDM is biocompatible and osteoinductive. Thus, PDDM which requires a partial demineralization process is an interesting point of research to be studied for its ability for contour augmentation in the esthetic zone.

DETAILED DESCRIPTION:
Dentin tooth can be classified into three groups according to the degree of demineralization undemineralized dentin (UDD), partially demineralized dentin matrix (PDDM) (70% decalcified) and demineralized dentin matrix (DDM). Some authors have shown that UDD is less effective in bone formation whereas other studies have shown that DDM is biocompatible and also osteoinductive, similar to demineralized bone matrix. Valdes concluded in their in vitro study that PDDM with large particle (1000µm) has much more bone regenerative activity in comparison to UDD. This could be explained because demineralization enhances the osteoinduction capacity of tooth material by exposing organic substances within the teeth to the surface, increasing porosity and surface area, and decreasing crystallinity . Nevertheless, some authors have reported successful bone regeneration applying UDD. UDD can be easily obtained from a dentin grinder, after disinfection and cleaning process. PDDM can be only obtained from the tooth after a partial demineralization process of the dentin. In any case, teeth must be free of restorations and caries, and endodontic teeth must be excluded.

However, several animal studies showed that demineralized dentin matrix (DDM) is not only biocompatible but also osteoinductive, similar to demineralized bone matrix. Dentin also contains some growth factors common to a bone, namely, insulin-like growth factor-II, bone morphogenetic protein (BMP), and transforming growth factor-beta. While APDDM has limited osteogenic potential but could be a suitable scaffold for osteoblastic cells. Furthermore, APDDM resists the rapid resorption of graft material. Complete resorption of DDM and remodeling into host bone has been reported to require >6 months. APDDM appears to resorb more slowly because it contains approximately 70% of original dentin matrix mineral. This partial demineralization of dentin matrix may affect the long-term stability of regenerated bone. While DDM may constitute an excellent BMP-2 carrier, APDDM could be a suitable substrate for cell attachment and differentiation. Notably, partial demineralization of dentin exposes collagen fiber, which enables cells to easily attach to substrate; the growth factors released from APDDM might concurrently stimulate osteoblastic differentiation. Furthermore, residual mineral in APDDM could enhance osteoclastic activity, thereby promoting bone remodeling. These factors may have contributed to the rapid and sufficient bone formation for dental implant placement with primary fixation.

To date, no other trial has been published that has used autogenous dentin as a graft material to resolve the periodontal defects on the distal aspect of the second molar derived from LTM extraction with post-operative clinical and CBCT monitoring. This present study was conducted to compare Early implant placement with Simultaneous Contour Augmentation using Partially demineralized dentin graft covered with a collagen membrane versus Early implant placement with Simultaneous Contour Augmentation using bovine xenograft covered with a collagen membrane in terms of esthetic and bone level changes during the first year of functional loading.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥20 years.
2. Mild smokers <1 pack of cigarettes a day
3. Capable of understanding or signing the informed consent form before surgery and capable of meeting oral cleaning requirements for implant placement
4. Healthy individuals with no systemic disease
5. Patients who have a single non-restorable tooth in the esthetic zone
6. Thin buccal plate of bone < 1mm prior to tooth extraction indicated for early implant placement with the ability to place a bone level implant able to achieve 35 N cm stability after placement.

Exclusion Criteria:

* 1) A habit of bruxism or inability to achieve requirements for oral cleaning 2) The presence of acute or chronic infection at the site of tooth extraction with lack of treatment for periodontal disease, or x-rays showing loss of alveolar bone on the adjacent teeth 3) Subjects who have a systemic disease which affects bone healing as diabetes and Paget's disease 4) Use of steroid therapy or under current treatment by chemotherapy or radiation therapy to the head and neck (as Bisphosphonates) 5) Pregnant or breastfeeding women

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Peri-implant soft tissue esthetics | After 3 months
  By probe measure Pink esthetic score from 0-10 for Mesial papilla, Distal papilla, Level of soft-tissue margin, Soft-tissue contour, Alveolar process and Color Texture

SECONDARY OUTCOMES:
Vertical buccal bone level changes | after 3 months of surgery
  by Cone beam computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: rana Sa Al Qahtani, master, Principal Investigator — research ethics committee , cairo university
Locations (1):
- Rana Saeed Al Qahtani, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided